CLINICAL TRIAL: NCT03126617
Title: Expanded Access to Elotuzumab (Empliciti) for Multiple Myeloma
Status: No longer available | Type: Expanded Access
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: EAP-01-CA204
Record Dates: First submitted 2017-04-18; First posted 2017-04-24 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: Elotuzumab — Elotuzumab (Emplicitii) is a Signaling Lymphocytic Activation Molecule Family member 7 (SLAMF7) directed immunostimulatory antibody approved by the US Food and Drug Administration (FDA) and indicated in combination with lenalidomide and dexamethasone for the treatment of patients with multiple myeloma who have received one to three prior therapies. Please contact your physician for more details.
  Other Names: Empliciti; BMS-901608

SUMMARY:
At BMS, we work with physicians/investigators to make investigational products available to patients with life-threatening diseases that have exhausted other treatment options and where there is a reasonable expectation of benefit over risk.

When contacted by a treating physician, BMS will consider requests for providing early patient access to Elotuzumab in patients with multiple myeloma who are residents of Belgium, Thailand, Turkey, Argentina, and Colombia.

DETAILED DESCRIPTION:
Choosing to participate in an early patient access program is an important personal decision. Talk with your doctor and family members or friends about deciding to participate in an early patient access program.

To learn more about early patient access programs, your doctor may contact BMS using the information provided below.

ELIGIBILITY:
Specific eligibility criteria must be met for access outside of a clinical trial.

These inclusion criteria include:

* The illness must be serious or life threatening
* There are no other viable options (including approved products or active clinical trials)
* There is sufficient evidence that the potential benefit to the patient would likely outweigh the potential risks based on what is known at the time
* Other defined inclusion/exclusion criteria could be applicable.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Information for Early Patient Access to Investigational Drugs — https://www.bms.com/healthcare-providers/early-patient-access-to-investigational-medicine.html